CLINICAL TRIAL: NCT07107529
Title: EFfIcacy and Tolerability of FIXed Duration Teclistamab and Talquetamab FOR FRAIL Patients With Newly Diagnosed Multiple Myeloma (2 Cohort Study) - the EMN 37 FITFIX FOR FRAIL Trial
Brief Title: Study for Frail Patients With Newly Diagnosed Multiple Myeloma Treated With Daratumumab With Teclistamab or Talquetamab.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: EMN Trial Office S.r.l. Impresa Sociale (Other); HOVON - Dutch Haemato-Oncology Association (Other); PETHEMA Foundation (Other); Nordic Myeloma Study Group (Other); Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN37; 2024-520433-76-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma (MM)
Keywords: Newly diagnosed multiple myeloma (NDMM); Frail patient; Talquetamab; Teclistamab
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Tec-Dara
  Interventions: Drug: Teclistamab; Drug: Daratumumab
- Cohort 2 (Experimental): Tal-Dara
  Interventions: Drug: Talquetamab; Drug: Daratumumab

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered via a subcutaneous injection (SC), fixed duration and will be retreated until disease progression or intolerable toxicity.
  Arms: Cohort 1
Drug: Talquetamab — Talquetamab will be administered via a subcutaneous injection (SC), fixed duration and will be retreated until disease progression or intolerable toxicity.
  Arms: Cohort 2
Drug: Daratumumab — Dartumumab will be administered via a subcutaneous injection (SC), fixed duration and will be retreated until disease progression or intolerable toxicity.

SUMMARY:
This is a multicenter, open-label phase II study with 2 parallel cohorts for frail patients with newly diagnosed multiple myeloma treated with daratumumab in combination with teclistamab and talquetamab.

The main purpose of this study is to determine the progression free survival at 18 months in patients treated with teclistamab and daratumumab (Cohort 1) or talquetamab and daratumumab (Cohort 2).

DETAILED DESCRIPTION:
This study will consist of 4 phases:

* Initial treatment phase where patients will receive fixed duration of Tec-Dara or Tal-Dara.
* TFI.
* Re-treatment phase, where patients with confirmed PD will continue treatment with Tec-Dara or Tal-Dara per their assignment in the initial treatment phase.
* Post-treatment follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age and capable of giving informed consent and must sign an informed consent form (ICF), indicating that they understand the purpose of, and procedures required for, the study and is willing to participate in the study
2. Newly diagnosed and treatment-naïve patients with a confirmed diagnosis of MM with measurable disease according to IMWG criteria
3. Measurable disease defined as M-protein in the serum (≥1 g/dL) or serum free light chain assay ≥10 mg/dL [≥100 mg/L] and abnormal serum immunoglobulin kappa/lambda FLC ratio
4. Frail according to the Simplified IMWG frailty index
5. Have clinical laboratory values meeting defined range
6. Patients of childbearing potential must agree to use adequate/highly effective contraception from the time of signing the informed consent form through 3 months after the last dose of study drug

Exclusion Criteria:

1. Non-secretory MM or measurable disease by urine or plasmacytoma only
2. Central nervous system involvement of myeloma
3. Significant pulmonary dysfunction
4. Stroke, transient ischemic attack, or seizure within 6 months of eligibility
5. Evidence of active systemic viral, fungal, or bacterial infections, requiring systemic antimicrobial therapy
6. HIV and Hepatitis infections
7. Exclude for any of the following:

   1. Any history of malignancy other than MM which is considered at high risk of recurrence requiring treatment or a malignancy that has been treated with chemotherapy currently affecting bone marrow capacity.
   2. Any active malignancy (ie, progressing or requiring treatment change in the last 24 months) other than multiple myeloma.
8. Active autoimmune disease requiring systemic immunosuppressive therapy within 6 months before eligibility
9. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study treatment or its excipients (refer to IB and most recently applicable RSI)
10. Extensive radiotherapy within 14 days or focal radiation only within 7 days of eligibility
11. Current or active therapy for multiple myeloma or received a cumulative dose corticosteroids equivalent to >40 mg dexamethasone within the 14 days prior to C1D1
12. Received a live attenuated vaccine ≤4 weeks before eligibility. Non-live vaccines or non-replicating authorized for emergency use (eg, COVID-19) are allowed
13. Received a strong CYP3A4 inducer or use of St. John's wort ≤5 half-lives prior to dosing
14. Patient had major surgery or significant traumatic injury within 2 weeks prior to eligibility. Kyphoplasty or Vertebroplasty is not considered major surgery
15. Have received an investigational drug (including investigation vaccines) or used an invasive investigational medical device <4 week or 5 PK half-lives, before eligibility or is currently enrolled in an interventional investigational study except if only long-term survival data are collected
16. Concurrent medical or psychiatric condition or disease (eg, uncontrolled diabetes, alcohol or drug abuse, severe dementia or altered mental status), that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participation in the study
17. Any other issue that would impair the ability of the patient to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (eg,, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per IMWG criteria | 18 months
  defined as the time from the date of randomization until the first occurrence of disease progression or death from any cause, whichever occurs earlier, where disease progression is determined per IMWG criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | 9 years
  Measured from the date of from randomization to the date the subject's death.
Minimal Residual Disease (MRD) negativity rate | 18 months
  Minimal Residual Disease (MRD) negative as determined by NGF at 10^-5 sensitivity level per International Myeloma Working Group (IMWG) criteria.
Minimal Residual Disease (MRD) negative CR | 18 months
  Minimal Residual Disease (MRD) negative Complete Remission (CR) at the end of fixed treatment duration status as determined by NGF at 10^-5 sensitivity level and who also achieve CR or better per International Myeloma Working Group (IMWG) criteria.
Sustained Minimal Residual Disease (MRD) negative CR | 9 years
  Sustained MRD-negative CR is defined as patients with CR or better who sustain MRD-negative status, as determined NGF at 10^-5.
IMWG best response | 18 months
  To evaluate the proportion of IMWG best response achieved by a patient during the study. Subject will be classified as Not Evaluable (NE) if they will not have any evaluable response assessment.
Time to response | 9 years
  Time from the date of randomization to the date of first documentation of a confirmed response (partial response) as per IMWG response criteria, for patients who have PR or better as their best response.
Time to best response | 9 years
  Time from the date of randomization to the date of first best response as per IMWG response criteria.
Event free survival (EFS) | 9 years
  Time from the date of randomization to the date of first documented disease progression, as defined in the IMWG criteria, or death due to any cause or treatment discontinuation due to toxicity, whichever occurs first.
Progression Free Survival 2 (PFS2) | 9 years
  Time from the randomization date to the date of event, which is defined as death from any cause or progression disease on the next line of therapy, whichever occurs first.
Time to Next Treatment (TNT) | 9 years
  Time from the randomization date to the date of event, which is defined as the start of the next line of therapy or death from any cause, whichever occurs first.
Adverse Events | 9 years
  Incidence and severity of Adverse Events during initial therapy, Treatment-Free-Interval (TFI) and after restarting therapy.
Discontinuation | 9 years
  Discontinuation rate and cause due to treatment related toxicity during initial therapy and after restarting therapy, including overall discontinuation rate, discontinuation rate of daratumumab, teclistamab and talquetamab.
Change from Baseline in Health-Related Quality of Life as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) Scale Score | Up to 9 years
  The EORTC QLQ-C30 includes 30 items in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single symptom items.
  The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.
Change from Baseline in Health-Related Quality of Life as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Myeloma 20 (EORTC-MY-20) Scale Score | Up to 9 years
  The EORTC-QLQ-MY20 is a specialised tool designed to assess the quality of life in myeloma patients.
  Scores are linearly transformed to a 0-100 scale, where higher scores on the symptom scales indicate worse outcomes.
Change from Baseline in Health-Related Quality of Life as Assessed by Activities of Daily Living (ADL) questionnaire | Up to 9 years
  The ADL questionnaire assesses functional status by measuring independence in six daily activities.
  The ADL scale is scored from 0 to 8, where higher scores indicate greater independence with daily activities.
Change from Baseline in Health-Related Quality of Life as Assessed by Instrumental Activities of Daily Living (IADL) questionnaire | Up to 9 years
  The IADL assesses instrumental activities of daily living, including telephone use, laundry, shopping, food preparation, and mode of transportation.
  The IADL scale is scored from 0 to 8, with higher scores indicating greater independence.
Change from Baseline in Health-Related Quality of Life as Assessed by Scale of Subjective Total Taste Acuity (STTA) | Up to 9 years
  The STTA scale assesses the taste acuity during treatment. The STTA scale is scored from 0 to 4, where 4 indicates almost complete loss of taste acuity.
Change from Baseline in the geriatric assessment as Assessed by Geriatric Depression Scale (GDS) | Up to 9 years
  The GDS scale assesses the depressive symptoms in frail elderly patients. The GDS scale is scored from 0 to 15. Score 1 point for each bolded answer. A score of 5 or more suggests depression.
Change from Baseline in the geriatric assessment as Assessed by Mini Nutritional Assessment (MNA) questionnaire | Up to 9 years
  The MNA is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition.
  The MNA scale is scored from 1 to 30. A higher score represents good nutrition, a score less then 17 represents malnutrition.
Change from Baseline in the geriatric assessment as Assessed by Mini-Mental State Examination (MMSE) | Up to 9 years
  The MMSE is an 11-question tool to assess mental status, testing five cognitive areas.
  The MMSE scale is scored from 1 to 30. A higher score represents good mental state.
Change from Baseline in the geriatric assessment as Assessed by Geriatric Assessment in Hematology (GAH) scale | Up to 9 years
  The GAH scale predicts treatment tolerability in older patients diagnosed with hematological malignancies.
  The 30-item GAH scale was designed through a multi-step process to cover 8 relevant dimensions. Higher scores indicate a more frail or vulnerable patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Zweegman, Principal Investigator — Vrije Universiteit Medical Center (VUMC); Maria-Victoria Mateos, Principal Investigator — University of Salamanca; Fredrik Schjesvold, Principal Investigator — Oslo University Hospital; Alessandra Larocca, Principal Investigator — A.O.U. Città della Salute e della Scienza di Torino; Niels van de Donk, Principal Investigator — Vrije Universiteit Medical Center (VUMC)

IPD SHARING:
Plan to Share IPD: No